CLINICAL TRIAL: NCT02982863
Title: Treatment Patterns of Newly Initiated Oral Anticoagulants on Japanese Non-valvular Atrial Fibrillation Patients Using a Japanese Claims Database
Brief Title: Treatment Pattern of Oral Anticoagulants (OAC) in Japan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0279
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- All Patients

SUMMARY:
1. To understand the treatment patterns of OACs and baseline patient characteristics of Japanese Non-Valvular Atrial Fibrillation (NVAF) patients
2. To determine whether warfarin and dabigatran new user group can be balanced using propensity score matching using pre-specified baseline covariates.
3. As an exploratory analysis, to assess mean duration of on-therapy follow-up time in database

ELIGIBILITY:
Inclusion criteria:

* Patients aged >18 year-old with confirmed diagnosis of NVAF (ICD 10 code I48), being new starters of either dabigatran, warfarin, apixaban or edoxaban, having no prescription of other OACs for12 months prior to the index date (defined as the first prescription of OACs (the period is defined as baseline period)), and having an index date between 14 Mar 2011 to 30 June 2016

Exclusion criteria:

* Patients having less than 12 months of enrolment prior to the index date , being dialysis or kidney transplant recipients in baseline period, having either atrial flutter, valvular AF, mechanical valve placement, rheumatic AF, and/or mitral valve prolapse/regurge/stenosis in baseline period, and having record of deep vein thrombosis or pulmonary embolism < 6 months before Atrial Fibrillation (AF) diagnosis in baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Data Vision (MDV) clinical database
Sampling Method: Non-Probability Sample
Enrollment: 48696 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- NISED Center, Tokyo, Shinagawa, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective, observational study using health insurance claims data.48696 patients were prescribed dabigatran, warfarin, apixaban, edoxaban, or rivaroxaban as the first OACs but 50 patients were removed as they took more than one these drugs. Thus only 48646 patients were prescribed the drugs of interest.
Pre-assignment Details: The Japanese patients diagnosed as Non-Valvular Atrial Fibrillation (NVAF) between April 2010 and June 2016, were prescribed dabigatran, warfarin, apixaban, edoxaban, or rivaroxaban as the first OACs.
  DPC; Diagnosis Procedure Combination (DPC)
Groups:
- Dabigatran: Patients prescribed dabigatran as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
- Warfarin: Patients prescribed warfarin as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
- Apixaban: Patients prescribed Apixaban as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
- Rivaroxaban: Patients prescribed Rivaroxaban as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
- Edoxaban: Patients prescribed Edoxaban as the first Oral Anticoagulants (OACs) with nonvalvular atrial fibrillation.
Period: Overall Study
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Started | 5745 | 16745 | 13238 | 10158 | 2760
Completed | 4936 | 12484 | 11386 | 8758 | 2268
Not Completed | 809 | 4261 | 1852 | 1400 | 492
Not completed — Not eligible patients | 809 | 4261 | 1852 | 1400 | 492

BASELINE CHARACTERISTICS:
Population: Eligible patient who were prescribed dabigatran, warfarin, apixaban, or edoxaban as the first OACs
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban | Total
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268 | 39832
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (10) | 78 (10) | 77 (10) | 74 (11) | 77 (10) | 76 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1625 | 5068 | 4737 | 3183 | 1130 | 15743
  Male | 3311 | 7416 | 6649 | 5575 | 1138 | 24089

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients by Each Type of Study-target OAC Drug Prescribed for New Users of Anticoagulants With NVAF
Description: Number of patients by each type of study-target OAC drug (dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban) prescribed as the first Oral Anticoagulants (OAC) with Non-valvular atrial fibrillation (NVAF)
Time Frame: Day 1
Population: Patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 5745 | 16745 | 13238 | 10158 | 2760
Participants | 4936 | 12484 | 11386 | 8758 | 2268

2. Primary Outcome: Number of Patients Prescribed OAC Drug Dabigatran by Dosage
Description: Number of patients prescribed OAC drug dabigatran at the index date by dosage. If a patient had more than one prescriptions of an OAC at the day, the patient was multiple-counted.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran
Number analyzed (Participants) | 4936
Participants
  75 milligram (mg) | 58
  110 mg | 164
  150 mg | 354
  220 mg | 3343
  225 mg | 5
  300 mg | 1072
  440 mg | 1

3. Primary Outcome: Number of Patients Prescribed OAC Drug Warfarin by Dosage
Description: Number of patients prescribed OAC drug Warfarin at the index date by dosage. If a patient had more than one prescriptions of an OAC at the day, the patient was multiple-counted.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin
Number analyzed (Participants) | 12484
Participants
  0.002 mg | 2
  0.006 mg | 1
  0.125 mg | 3
  0.2 mg | 4
  0.25 mg | 338
  0.3 mg | 2
  0.374 mg | 1
  0.5 mg | 1726
  0.6 mg | 3
  0.625 mg | 2
  0.65 mg | 1
  0.7 mg | 1
  0.75 mg | 256
  0.8 mg | 1
  0.875 mg | 3
  0.9 mg | 2
  1 mg | 3125
  1.2 mg | 2
  1.25 mg | 62
  1.3 mg | 1
  1.5 mg | 630
  1.55 mg | 1
  1.7 mg | 2
  1.75 mg | 66
  1.8 mg | 2
  1.9 mg | 1
  2 mg | 4711
  2.2 mg | 1
  2.25 mg | 54
  2.3 mg | 1
  2.4 mg | 3
  2.5 mg | 462
  2.7 mg | 1
  2.75 mg | 24
  3 mg | 1913
  3.2 mg | 1
  3.25 mg | 17
  3.3 mg | 1
  3.5 mg | 128
  3.7 mg | 1
  3.75 mg | 9
  4 mg | 421
  4.25 mg | 3
  4.5 mg | 41
  4.6 mg | 1
  4.75 mg | 1
  5 mg | 468
  5.5 mg | 9
  6 mg | 25
  6.5 mg | 2
  7 mg | 8
  7.75 mg | 1
  8 mg | 3
  9 mg | 1
  10 mg | 16
  17.5 mg | 1
  20 mg | 3
  30 mg | 12
  40 mg | 3
  50 mg | 1

4. Primary Outcome: Number of Patients Prescribed OAC Drug Rivaroxaban by Dosage
Description: Number of patients prescribed OAC drug rivaroxaban at the index date by dosage. If a patient had more than one prescriptions of an OAC at the day, the patient was multiple-counted.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 8758
Participants
  5 mg | 14
  7.5 mg | 3
  9.9 mg | 3
  9.99 mg | 2
  10 mg | 4372
  10.005 mg | 4
  10.05 mg | 10
  10.5 mg | 1
  15 mg | 4340
  20 mg | 5
  22.5 mg | 1
  30 mg | 72

5. Primary Outcome: Number of Patients Prescribed OAC Drug Apixaban by Dosage
Description: Number of patients prescribed OAC drug Apixaban at the index date by dosage. If a patient had more than one prescriptions of an OAC at the day, the patient was multiple-counted.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban
Number analyzed (Participants) | 11386
Participants
  1.25 mg | 2
  2.5 mg | 428
  3.75 mg | 2
  5 mg | 6300
  7.5 mg | 1
  10 mg | 4789
  15 mg | 1
  20 mg | 27
  25 mg | 2
  35 mg | 1

6. Primary Outcome: Number of Patients Prescribed OAC Drug Edoxaban by Dosage
Description: Number of patients prescribed OAC drug edoxaban at the index date by dosage. If a patient had more than one prescriptions of an OAC at the day, the patient was multiple-counted.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban
Number analyzed (Participants) | 2268
Participants
  15 mg | 279
  30 mg | 1594
  60 mg | 412

7. Secondary Outcome: Baseline Characteristics: Age
Description: Baseline characteristics of patients in each treatment group: age
Time Frame: 1 day
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Years | 72 (10) | 78 (10) | 77 (10) | 74 (11) | 77 (10)

8. Secondary Outcome: Baseline Characteristics: Gender
Description: Baseline characteristics of patients in each treatment group: gender
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  Female | 1625 | 5068 | 4737 | 3183 | 1130
  Male | 3311 | 7416 | 6649 | 5575 | 1138

9. Secondary Outcome: Baseline Characteristics: Year of Initiating Treatment
Description: Baseline characteristics of patients in each treatment group: year of initiating treatment
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  2011/3/14-2012/2/29 | 404 | 1138 | 0 | 0 | 8
  2012/3/1-2013/2/28 | 1259 | 2002 | 0 | 175 | 32
  2013/3/1-2014/2/28 | 1081 | 2292 | 188 | 1868 | 29
  2014/3/1-2015/2/28 | 1019 | 2808 | 3455 | 2182 | 158
  2015/3/1-2016/2/29 | 919 | 3217 | 5634 | 3302 | 1289
  2016/3/1-2016/6/30 | 254 | 1027 | 2109 | 1231 | 752

10. Secondary Outcome: Baseline Characteristics: Speciality of Prescribers of OAC
Description: Baseline characteristics of patients in each treatment group: speciality of prescribers of OAC.
  int.= internal; Med.= Medicine
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  Internal medicine | 1689 | 4316 | 3943 | 2816 | 654
  Psychodiagnosis medical | 2 | 3 | 2 | 1 | 1
  Psychiatry | 9 | 38 | 30 | 20 | 7
  Neurology | 0 | 1 | 7 | 3 | 2
  Respiratory | 66 | 180 | 95 | 72 | 17
  Gastroenterology | 106 | 283 | 100 | 125 | 26
  Cardiology | 1457 | 2447 | 2610 | 2268 | 465
  Allergy | 1 | 9 | 1 | 0 | 0
  Rheumatology | 7 | 11 | 6 | 3 | 2
  Pediatrics | 0 | 5 | 4 | 4 | 0
  Surgery | 109 | 514 | 202 | 175 | 52
  Orthopedics | 113 | 550 | 212 | 178 | 317
  Plastic surgery | 5 | 21 | 10 | 5 | 2
  Cranial nerve surgery | 319 | 668 | 932 | 654 | 164
  Thoracic surgery | 10 | 58 | 27 | 25 | 3
  Cardiovascular surgery | 87 | 405 | 115 | 147 | 54
  Pediatric surgery | 0 | 0 | 1 | 0 | 0
  Obstetrics and gynecology | 4 | 11 | 9 | 5 | 6
  Ophthalmology | 19 | 38 | 26 | 36 | 5
  Otorhinolaryngology | 8 | 47 | 25 | 19 | 5
  Rehabilitation | 30 | 127 | 86 | 86 | 12
  Radiology | 4 | 12 | 8 | 5 | 0
  Neuropathic internal medicine | 210 | 410 | 518 | 415 | 74
  Gastrointestinal | 0 | 17 | 5 | 3 | 1
  Dermatology | 9 | 41 | 23 | 23 | 3
  Urology | 31 | 161 | 76 | 55 | 15
  Gynecology | 2 | 2 | 1 | 2 | 0
  Respiratory medicine | 36 | 161 | 112 | 75 | 18
  Cardiovascular internal medicine | 444 | 1258 | 1930 | 1218 | 301
  Diabetes | 3 | 14 | 8 | 10 | 0
  Nephrology | 13 | 85 | 27 | 15 | 7
  Hemodialysis | 1 | 8 | 0 | 0 | 0
  Metabolism internal medicine | 0 | 3 | 4 | 7 | 0
  Endocrinology | 8 | 24 | 16 | 15 | 2
  Emergency medicine | 18 | 59 | 54 | 46 | 11
  Gastroenterological medicine | 53 | 270 | 61 | 85 | 20
  Digestive surgery | 6 | 25 | 7 | 10 | 4
  Hepato-biliarypancreatic surgery | 0 | 4 | 4 | 1 | 1
  Diabetes medicine | 4 | 19 | 12 | 9 | 0
  Large intestine and proctology | 0 | 1 | 0 | 0 | 0
  Connective tissue disease & iheumatic int. med. | 2 | 8 | 1 | 1 | 0
  Stroke | 2 | 6 | 5 | 0 | 0
  Oncotherapy | 2 | 6 | 0 | 1 | 1
  Comprehensive medical care | 13 | 56 | 12 | 9 | 3
  Breast and thyroid surgery | 0 | 3 | 0 | 2 | 1
  Pediatric cardiology | 0 | 3 | 0 | 0 | 0
  Palliative care | 0 | 1 | 0 | 0 | 0
  Hematology & medical Oncology | 0 | 1 | 1 | 1 | 1
  Psychiatry & neurology | 0 | 0 | 1 | 0 | 0
  Endocrinology & metabolism | 1 | 1 | 2 | 1 | 0
  Unknown | 27 | 59 | 38 | 83 | 8
  Hematology | 6 | 27 | 11 | 20 | 2
  Anesthesiology | 0 | 7 | 6 | 4 | 1

11. Secondary Outcome: Baseline Characteristics: History of Disease
Description: Baseline characteristics of patients in each treatment group: history of disease and hospitalization.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  Stroke or transient ischemic attack | 63 | 145 | 128 | 85 | 21
  Myocardial infarction | 317 | 903 | 890 | 629 | 178
  Coronary artery disease | 39 | 87 | 79 | 53 | 25
  Heart failure | 1899 | 6750 | 5099 | 3580 | 977
  Diabetes mellitus | 1979 | 4804 | 4255 | 3324 | 841
  Dyslipidemia | 1366 | 2888 | 3109 | 2402 | 597
  Arterial hypertension | 2938 | 8501 | 6990 | 5357 | 1344
  Peripheral artery disease | 580 | 1538 | 1290 | 933 | 252
  Peptic ulcer disease | 958 | 2301 | 2148 | 1558 | 452
  Dementia | 107 | 447 | 348 | 268 | 90
  Malignant lymphoma | 62 | 171 | 159 | 109 | 41
  Leukemia | 34 | 161 | 107 | 82 | 27
  Solid tumor cancer | 1501 | 3830 | 3413 | 2524 | 678
  Kidney impairment | 199 | 697 | 527 | 360 | 118
  Liver disease | 784 | 1777 | 1576 | 1257 | 339
  Valvular disease | 1659 | 4294 | 2961 | 2561 | 615
  Bleeding (gastrointestinal, etc.) | 1619 | 3867 | 3567 | 2677 | 782

12. Secondary Outcome: Baseline Characteristics: History of Hospitalization
Description: Baseline characteristics: history of hospitalization
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants | 2384 | 9494 | 6517 | 4589 | 1412

13. Secondary Outcome: Baseline Characteristics: AF Risk Score
Description: Baseline characteristics of patients in each treatment group: Atrial Fibrillation (AF) risk score
  CHADS2: Congestive heart failure, Hypertension, Age, Diabetes, Stroke(doubled). CHADS2 score range from 0-6, with higher scores indicating the higher risk
  CHA2DS2VASc: Cardiac failure or dysfunction, Hypertension, Age 75 (doubled), Diabetes, Stroke (doubled) Vascular disease, Age 65-74 and Sex category (female) score. CHA2DS2VASc score range from 1-9, with higher scores indicating the higher risk.
  HAS-BLED: Hypertension, Abnormal renal function, Abnormal hepatic function. HAS-BLED score range from 0-8, with higher scores indicating the higher risk.
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  0 (CHADS2) | 707 | 750 | 1150 | 1072 | 238
  1 (CHADS2) | 1103 | 2239 | 2504 | 1928 | 513
  2 (CHADS2) | 1131 | 2816 | 2330 | 2022 | 517
  3 (CHADS2) | 1053 | 3458 | 2787 | 2005 | 523
  4 (CHADS2) | 582 | 1897 | 1611 | 1014 | 267
  5 (CHADS2) | 243 | 816 | 626 | 459 | 125
  6 (CHADS2) | 117 | 508 | 378 | 258 | 85
  0 (CHA2DS2VASc) | 198 | 182 | 280 | 295 | 66
  1 (CHA2DS2VASc) | 547 | 585 | 773 | 783 | 140
  2 (CHA2DS2VASc) | 878 | 1500 | 1692 | 1481 | 305
  3 (CHA2DS2VASc) | 968 | 2380 | 2213 | 1735 | 497
  4 (CHA2DS2VASc) | 916 | 2685 | 2216 | 1718 | 432
  5 (CHA2DS2VASc) | 690 | 2496 | 2070 | 1348 | 380
  6 (CHA2DS2VASc) | 441 | 1482 | 1165 | 769 | 241
  7 (CHA2DS2VASc) | 188 | 738 | 644 | 402 | 129
  8 (CHA2DS2VASc) | 96 | 369 | 257 | 188 | 61
  9 (CHA2DS2VASc) | 14 | 67 | 76 | 39 | 17
  0 (HAS-BLED) | 297 | 245 | 422 | 432 | 68
  1 (HAS-BLED) | 1276 | 2303 | 2848 | 2228 | 545
  2 (HAS-BLED) | 1616 | 4180 | 3725 | 2884 | 746
  3 (HAS-BLED) | 1192 | 3738 | 2837 | 2159 | 590
  4 (HAS-BLED) | 458 | 1562 | 1258 | 872 | 270
  5 (HAS-BLED) | 89 | 403 | 266 | 162 | 46
  6 (HAS-BLED) | 7 | 53 | 30 | 20 | 3
  7 (HAS-BLED) | 1 | 0 | 0 | 1 | 0
  8 (HAS-BLED) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Baseline Characteristics: Concomitant Medication
Description: Baseline characteristics of patients in each treatment group:
  concomitant medication
Time Frame: Day 1
Population: eligible patients prescribed dabigatran, warfarin, apixaban, rivaroxaban, or edoxaban as the first OAC
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Number analyzed (Participants) | 4936 | 12484 | 11386 | 8758 | 2268
Participants
  Aspirin | 989 | 2848 | 2027 | 1621 | 377
  Ticlodipine | 69 | 179 | 115 | 95 | 12
  Cilostazole | 199 | 522 | 466 | 306 | 66
  Clopidogrel | 346 | 1049 | 1031 | 767 | 153
  ARB or ACE | 1649 | 4773 | 3650 | 2954 | 661
  Beta blocker | 1779 | 4376 | 4272 | 3137 | 768
  Amiodarone | 62 | 388 | 301 | 138 | 31
  Procainamide | 14 | 40 | 43 | 17 | 8
  Disopyramide | 102 | 230 | 180 | 150 | 34
  Flecainide | 130 | 105 | 237 | 150 | 33
  Pilsicainide | 582 | 726 | 970 | 885 | 145
  Calcium channel blockers (CCB) | 2176 | 5755 | 5148 | 3955 | 955
  Digoxin | 506 | 1959 | 944 | 896 | 134
  Diuretics | 1277 | 5901 | 3698 | 2480 | 681
  Statins | 1029 | 2736 | 2364 | 1876 | 407
  Proton pump inhibitor | 1869 | 5512 | 4583 | 3506 | 970
  H2 receptor antagonist | 761 | 2559 | 1673 | 1365 | 367

ADVERSE EVENTS:
Description: The outcomes of the study were the baseline characteristics (pre-treatment) and medication prescriptions. The study was not desinged to assess adverse event; therefore safety reporting was not applicable for this study.
Arm/Group | Dabigatran | Warfarin | Apixaban | Rivaroxaban | Edoxaban
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Generalizability of findings may be limited outside of population. The data in Medical Data Vision Co., Ltd. (MDV) database is collected from DPC hospitals that may contain out-patient data with greater disease severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes